CLINICAL TRIAL: NCT02763904
Title: Systematic Oral Nutritional Support in Hospitalized, Moderately Hypophagic Patients At Nutritional Risk Receiving Dietary Counseling: a Randomized, Controlled Trial
Brief Title: Systematic Oral Nutritional Support in Hospitalized, Moderately Hypophagic Patients At Nutritional Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emanuele Cereda (Other)
Responsible Party: Sponsor-Investigator, Emanuele Cereda, Fondazione IRCCS Policlinico San Matteo di Pavia, Fondazione IRCCS Policlinico San Matteo di Pavia
Organization: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150005564
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Nutritional Support
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive nutritional counseling (Experimental): Dietary counseling + energy dense oral nutritional supplements
  Interventions: Dietary Supplement: Intensive nutritional counseling
- Dietary counseling (Active Comparator): Dietary counseling
  Interventions: Other: Dietary counseling

INTERVENTIONS:
Dietary Supplement: Intensive nutritional counseling — Dietary counseling + energy-dense oral nutritional supplements since admission
  Arms: Intensive nutritional counseling
Other: Dietary counseling — Dietary counseling alone. In case of inadequate energy intake patients will receive oral nutritional supplements since day 8 from admission (after the evaluation of the primary end point)
  Arms: Dietary counseling

SUMMARY:
Protein-calorie malnutrition is a frequent comorbidity in hospitalized patients and there is evidence that the nutritional status may influence the response to drug treatment, mortality, susceptibility to infections, the patient's functional status, duration of hospital stay and, consequently, overall healthcare costs. The causes of malnutrition are manifold. The underlying disease may in fact lead to an increase in the patient's energy needs, whether or not associated with a reduction in caloric intake. The same therapeutic treatments can further worsen the energy balance without considering that the patient can be kept fasting for the execution of some diagnostic procedures. Therefore, a further deterioration of nutritional status during hospitalization could occur.

International guidelines underline the utility to set a nutritional support whenever this is necessary, not only to prevent or treat malnutrition but also improve clinical outcomes. In this perspective, the improvement of oral diet and the use of oral nutritional supplements (ONS) represent the first-line strategy of intervention. Previous studies have shown that nutritional counseling, with or without the use of ONS, in patients with chronic disease is able to improve the calorie-protein intake, prevent deterioration of nutritional status, as well as to increase to a certain extent body weight. Particularly, energy-dense are more effective in increase energy intake. These data have highlighted the importance of a proper evaluation of the nutritional status of early detection of patients who could benefit of nutritional support. However, the independent role of the ONS in improving clinical outcome still needs to be established.

ELIGIBILITY:
Inclusion Criteria:

* Nutritional Risk Score [NRS-2002] ≥3
* assessed within 48 hours since admission
* expected length of stay ≥7 days
* written informed consent

Exclusion Criteria:

* age < 18 years
* ongoing or indication to artificial nutrition
* severe hypophagia (intake <50% of estimated requirements)
* scheduled for surgery
* indication to fasting
* physician-based contra-indication to use of liquid oral nutritional supplements (vomitus, severe nausea, diarrhea, dysphagia)
* physician-based indication to the of disease-specific oral nutritional supplements (e.g. kidney failure or pressure ulcers)
* terminal illness
* unavailability to planned measurements

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-07-30 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Body composition | 7 days
  Change in phase angle as assessed by vectorial impedance analysis

SECONDARY OUTCOMES:
Body composition | 14 days
  Change in phase angle as assessed by vectorial impedance analysis
Body composition | Hospital stay, an average of 17 days
  Change in phase angle as assessed by vectorial impedance analysis
Functional status | 7 days
  Change in handgrip strength as assessed by dynamometry
Functional status | 14 days
  Change in handgrip strength as assessed by dynamometry
Functional status | Hospital stay, an average of 17 days
  Change in handgrip strength as assessed by dynamometry
Energy intake | 7 days
  Protein-calorie intake as assessed by serial 24-hour dietary recall
Energy intake | 14 days
  Protein-calorie intake as assessed by serial 24-hour dietary recall
Infections | Hospital stay, an average of 17 days
  Incidence of new infections during the hospital stay
Adverse events | Hospital stay, an average of 17 days
  Gastrointestinal intolerance events

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Cereda, MD, PhD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo; Riccardo Caccialanza, MD, Study Chair — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Nutrition and Dietetics Service, Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided